CLINICAL TRIAL: NCT06968117
Title: Exploration of Pregnant Women's Reluctance Toward COVID-19 Vaccination
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0025_MATERNITE
Record Dates: First submitted 2025-05-12; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Vaccinate Against Covid-19; Reluctance Pregnant Women's

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women participating in the study on COVID-19 vaccination hesitancy.: This group consists of pregnant women, recruited during prenatal consultations, hospital admissions, or visits to obstetric emergencies. The aim is to explore their perceptions and hesitations regarding COVID-19 vaccination.

SUMMARY:
This study aims to explore the reasons behind the reluctance of pregnant women to get vaccinated against COVID-19. With the ongoing pandemic, it has become essential to understand the concerns that women have regarding the COVID-19 vaccine, especially during pregnancy. Pregnant women are at a higher risk of severe complications from COVID-19, including premature birth, preeclampsia, and the need for intensive care.The goal of this research is to identify the barriers that prevent pregnant women from getting vaccinated, whether they are based on fears, misconceptions, or a lack of information. By understanding these concerns, healthcare providers can have better conversations with their patients and provide accurate, evidence-based information to help them make informed decisions about their health and the health of their unborn child.Through interviews and visual methods, the study seeks to gather valuable insights into the emotional and psychological aspects of vaccine hesitancy among pregnant women. These findings will help develop a tool to assist healthcare providers in addressing vaccine hesitancy effectively, ensuring that women are given all the necessary information to make the best decision for their health and the well-being of their baby.

ELIGIBILITY:
Inclusion Criteria:

* During pregnancy follow-up consultations,
* Following their visit to the Gynecology-Obstetrics emergency department, regardless of the reason,
* Hospitalized in the diabetology department or in the high-risk pregnancy (HRP) or postpartum care department.

Exclusion Criteria:

* The patient is over 18 years old

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study participants will be selected from pregnant women attending pregnancy follow-up consultations, those who have visited the Gynecology-Obstetrics emergency department for any reason, and those hospitalized in the diabetes or high-risk pregnancy (GHR) departments or in postpartum care services. Participants must be over 18 years old and able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
The rate of vaccine hesitancy among pregnant women, assessed through a standardized questionnaire. | January 2021-April 2023

CONTACTS AND LOCATIONS:
Locations (1):
- France, Gonesse, France